CLINICAL TRIAL: NCT07240129
Title: Effect of Graded Motor Imagery on Shoulder Dysfunction Post Mastectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Abdallah Mohamed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005749
Record Dates: First submitted 2025-06-26; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Dysfunction
Keywords: Graded Motor Imagery; Post Mastectomy

STUDY DESIGN:
Intervention Model Description: Design of the study:
  In this study the patients will be randomly assigned into two equal groups (27 patients for each group)
Who Masked: Participant
Masking Description: Singl blind (participants)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (study group) (Active Comparator): This group includes 27 patients who will receive graded motor imagery (GMI) along with the conventional physiotherapy (It will include exercise like codman's pendulum exercises in flexion-extension, abduction-adduction, and circular motion, active assisted ROM exercises with a wand, capsular stretching, wall ladder, and shoulder wheel exercises). GMI is consists of a three-step process. Each step of will be carried out for two weeks, for 30 minutes on two separate days, for total 6 weeks
  Interventions: Other: Graded Motor Imagery (GMI); Other: Physical therapy program
- Group B (control group) (Placebo Comparator): This group includes 27 patients who will receive conventional physiotherapy treatment for improving ROM and decreasing pain. It will include exercise like codman's pendulum exercises in flexion-extension, abduction-adduction, and circular motion, active assisted ROM exercises with a wand, capsular stretching, wall ladder, and shoulder wheel exercises, 2 times / week for 6 weeks
  Interventions: Other: Physical therapy program

INTERVENTIONS:
Other: Graded Motor Imagery (GMI) — 1. Left/right judgements:
     It includes left/right judgments of photographs that depict the affected area.
  2. Imagined movements:
     Movement visualizations will be performed.
  3. Mirror therapy:
  It includes observation of the movements of unaffected body part in the mirror, 2 times / week for 6 weeks.
  Arms: Group A (study group)
Other: Physical therapy program — It will include exercise like codman's pendulum exercises in flexion-extension, abduction-adduction, and circular motion, active assisted ROM exercises with a wand, capsular stretching, wall ladder, and shoulder wheel exercises, 2 times / week for 6 weeks.
  Other Names: A group of exercises

SUMMARY:
One of the most common complications after breast cancer surgery is a functional limitation of the upper body. Up to 67% of breast cancer patients experience arm or shoulder impairment, including pain, numbness, loss of strength, and reduced ROM, after surgery.

Graded motor imagery is effective in reducing pain interference with function using a graded sequence of strategies including left/right judgements (implicit motor imagery), imagined movements (explicit motor imagery) and mirror therapy.

DETAILED DESCRIPTION:
54 female patients who have shoulder dysfunction post-mastectomy will participate in this study. Their ages will be ranged 35 to 55 years.

In this study the patients will be randomly assigned into two equal groups (27 patients for each group):

1. Group A (study group):

   This group includes 27 patients who will receive graded motor imagery (GMI) along with the conventional physiotherapy (It will include exercise like codman's pendulum exercises in flexion-extension, abduction-adduction, and circular motion, active assisted ROM exercises with a wand, capsular stretching, wall ladder, and shoulder wheel exercises). GMI is consists of a three-step process. Each step of will be carried out for two weeks, for 30 minutes on two separate days, for total 6 weeks.
2. Group B (control group):

This group includes 27 patients who will receive conventional physiotherapy treatment for improving ROM and decreasing pain. It will include exercise like codman's pendulum exercises in flexion-extension, abduction-adduction, and circular motion, active assisted ROM exercises with a wand, capsular stretching, wall ladder, and shoulder wheel exercises, 2 times / week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 35 to 55 years.
* All patients are post-mastectomized unilaterally.
* Female patients only.
* Patients have shoulder ROM restriction.
* Patients have shoulder pain more than 3 months (chronic).
* After 3 months post-surgery.

Exclusion Criteria:

* Having double mastectomy.
* Psychopathological disorders.
* Having other orthopedic problems (e.g. tendinitis, dislocation, osteoarthritis, referred pain to shoulder).
* Motor problems (e.g. tremor, dyskinesia).
* Metastasis.
* Visual impairment such that they could not read unaided or with their reading glasses.
* Having previously received GMI treatment.
* Diabetes mellitus.
* Having neurological problems as hemiplegia.
* Patients with lymphedema

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility is based on biological gender
Enrollment: 54 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Digital goniometer | From baseline to 6 weeks
  A device which measures joint ranges.
Handgrip dynamometer | From baseline to 6 weeks
  A valid tool for measuring handgrip strength in kilograms that provides an objective overview of upper limb functional integrity

SECONDARY OUTCOMES:
Visual analog scale | From baseline to 6 weeks
  A validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 means "no pain" and 10 means "worst pain."
Shoulder Pain and Disability Index | From baseline to 6 weeks
  Is a self-administered questionnaire that aims to measure pain and disability associated with shoulder disease with lower scores indicate little pain or disability and higher scores indicate higher pain and disability

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Abdallah, PhD, Principal Investigator — Teaching assistant of physical therapy for surgery, cairo university, egypt
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No